CLINICAL TRIAL: NCT05629039
Title: Volitional Help Sheet to Promote Smoking Cessation Among Young Adults in Indonesia
Brief Title: Implementing an Intervention Named Volitional Help Sheets to Reduce Smoking Behaviour Among Young Adults in Indonesia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manchester (Other)
Responsible Party: Principal Investigator, Rina Rahmatika, PhD Student, University of Manchester
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: VHS-Indonesia
Record Dates: First submitted 2022-09-22; First posted 2022-11-29 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Smoking Cessation
Keywords: Volitional help sheets; Young adults; Smoking cessation; Indonesia
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (10):
- Wave 1-Experimental Group (Experimental): The experimental group in Wave 1 will complete the baseline questionnaires (the socio-demographic, FTND, and COM-B questionnaires) followed by both the if-then list and the if-then link from the Volitional-Help Sheet as manipulations. The if-then list consists of several situations and solutions linked to smoking uptake in the volitional help sheet and the group will be informed that the activity will help to stop smoking. In addition, the if-then link consists of the situations in which people are urged to smoke and then link them to solutions that are most likely to help them abstain from starting smoking
  Interventions: Behavioral: Volitional Help Sheets
- Wave 1-Control Group (No Intervention): The control group participants will complete the baseline questionnaires (the socio-demographic questionnaire, the FTND, and the COM-B Questionnaire) without further intervention
- Wave 2-Control group (No Intervention): This group will complete the one-month follow-up questionnaires (the socio-demographic questionnaire, the FTND, and the COM-B Questionnaire) without further intervention
- Wave 2-Delayed VHS Group (Experimental): This group will receive the (delayed) Volitional Help Sheets intervention after completing the one-month follow-up questionnaires (the socio-demographic questionnaire, the FTND, and the COM-B Questionnaire).
  Interventions: Behavioral: Volitional Help Sheets
- Wave 2-Early VHS Group (Experimental): This group will complete the one-month follow-up questionnaires (the socio-demographic questionnaire, the FTND, and the COM-B Questionnaire) without further intervention
  Interventions: Behavioral: Volitional Help Sheets
- Wave 2-Repeated VHS group (Experimental): This group will complete the one-month follow-up questionnaires (the socio-demographic questionnaire, the FTND, and the COM-B Questionnaire), and receive a repeated, booster VHS intervention.
  Interventions: Behavioral: Volitional Help Sheets
- Wave 3-Control Group (No Intervention): This group will complete the six-month follow-up questionnaires. Due to ethical consideration, in wave three the control group will be offered the opportunity to complete the VHS form after they complete the follow-up assessments and the scores will not be included in the analysis.
- Wave 3-Delayed VHS Group (Experimental): This group will complete the six-month follow-up questionnaires (the socio-demographic questionnaire, the FTND, and the COM-B Questionnaire) without further intervention
  Interventions: Behavioral: Volitional Help Sheets
- Wave 3-Early VHS Group (Experimental): This group will complete the six-month follow-up questionnaires (the socio-demographic questionnaire, the FTND, and the COM-B Questionnaire) without further intervention
  Interventions: Behavioral: Volitional Help Sheets
- Wave 3-Repeated VHS Group (Experimental): This group will complete the six-month follow-up questionnaires (the socio-demographic questionnaire, the FTND, and the COM-B Questionnaire) without further intervention
  Interventions: Behavioral: Volitional Help Sheets

INTERVENTIONS:
Behavioral: Volitional Help Sheets — The volitional help sheet is an intervention which provides an opportunity for people to actively plan their behavioural changes by using a list of situations and solutions. The list of situations are critical situations which provoke unwanted behaviour, and the solutions are the responses to overcome the situations which urge the unexpected behaviour. In the context of smoking behaviour, the list of situations is the situations that will provoke cigarette uptake and the list of solutions is the appropriate responses to reduce or stop the urge to smoke.
  Other Names: Volitional help sheets for smoking cessation
  Arms: Wave 1-Experimental Group; Wave 2-Delayed VHS Group; Wave 2-Early VHS Group; Wave 2-Repeated VHS group; Wave 3-Delayed VHS Group; Wave 3-Early VHS Group; Wave 3-Repeated VHS Group

SUMMARY:
Indonesia is one of the countries that does not sign The World Health Organization Framework Convention on Tobacco Control (WHO-FCTC), and the numbers of Indonesian smokers increase every year. The Volitional-Help Sheet (VHS) has been used successfully to help people quit smoking, but has not yet been tested in Indonesia. The present study aims to adapt and implement the VHS to promote smoking cessation among smokers aged 20- 45 years. The main outcome measure is smoking abstinence; secondary outcomes are nicotine dependence, and capabilities, opportunities and motivations.

DETAILED DESCRIPTION:
The main outcome measure is smoking abstinence; secondary outcomes are nicotine dependence, and capabilities, opportunities and motivations. All participants will be smokers aged 20-45 years who will complete self-report measures of outcomes over three waves of data collection. Once baseline measures are collected, participants will be randomised at wave 1 to intervention versus control condition. Participants in the intervention group will complete the VHS for smoking cessation in addition to the baseline measures. At wave 2, one-month following wave 1, participants will again be randomised to intervention (complete the VHS) and control condition. There will thus be four conditions: control, early intervention, late intervention and repeated intervention. Outcomes will be assessed at wave 3, six-months after wave 2.

ELIGIBILITY:
Inclusion Criteria:

* Smokers whose ages are 20-45 years old

Exclusion Criteria:

* Non-smokers whose ages are below 20 years old and above 45 years old

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2700 (Estimated)
Dates: Start 2023-05-15 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Smoking Cessation | 6 months
  Participants will complete a self-report questionnaire to assess their cigarette uptake by ticking one of the following options: (a) I have never smoked (b) I have only tried smoking once (c) I used to smoke sometimes, but I never smoke cigarettes now (d) I sometimes smoke cigarettes now, but I do not smoke as many as one a week (e) I usually smoke between one and six cigarettes a week (f) I usually smoke more than six cigarettes a week. The code for the response of options "a-d" is 0, and "e-f" is 1.

SECONDARY OUTCOMES:
Nicotine dependence | 6 months
  The Fagerstrom nicotine dependence scale will assess nicotine dependence. The scoring method in FTND is 0 to 1 for yes/no items and a score of 0 to 3 for the multiple-choice items. The items are summed to yield a total score of 0-10. The higher the total FTND score, the more intense the smoker's physical dependence on nicotine.
Intervention evaluation | 6 months
  The Capability Opportunity Motivation-Behaviour (COM-B) Questionnaire will measure how the intervention contributes to the behaviour changes. The higher the score, the more the intervention contributes to the behaviour changes.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Armitage, Principal Investigator — University of Manchester; Tim Millar, Principal Investigator — University of Manchester
Locations (1):
- Rina Rahmatika, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No
The research team will receive anonymous data from the survey panel company. Therefore, there will be no identifiable data to be shared with other researchers.